CLINICAL TRIAL: NCT03098550
Title: Phase 1/2 Study to Evaluate the Safety and Preliminary Efficacy of Nivolumab Combined With Daratumumab in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Test the Safety and Effectiveness of Nivolumab Combined With Daratumumab in Patients With Pancreatic, Non-Small Cell Lung or Triple Negative Breast Cancers, That Have Advanced or Have Spread
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9GW; 2017-000367-33 (EudraCT Number)
Record Dates: First submitted 2017-03-28; First posted 2017-03-31 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Advanced Cancer
Keywords: Non-small cell lung cancer (NSCLC); Triple Negative Breast Cancer (TNBC); Pancreatic Cancer (PAC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Pancreatic Neoplasms | interventions — Nivolumab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immunotherapy Combination (Experimental): TNBC and PAC participants who are deriving clinical benefit will continue to be treated with the nivolumab plus daratumumab combination therapy
  Interventions: Biological: Nivolumab; Biological: Daratumumab
- Nivolumab Monotherapy (Experimental): NSCLC patients who are deriving clinical benefit will be treated with nivolumab monotherapy
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
Biological: Daratumumab — Specified dose on specified days
  Arms: Immunotherapy Combination

SUMMARY:
The purpose of this study is to determine whether a combination of Nivolumab and Daratumumab is safe and effective when treating Pancreatic, Non-Small Cell Lung or Triple Negative Breast Cancers, that have advanced or have spread.

ELIGIBILITY:
Inclusion Criteria:

For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

* Patients with metastatic or advanced solid tumors
* Women with histologically or cytologically confirmed triple negative breast carcinoma
* Participants with histologically or cytologically confirmed pancreatic adenocarcinoma
* Participants with histologically or cytologically confirmed Non Small Cell Lung Cancer (NSCLC)

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases.
* Any serious or uncontrolled medical disorder
* Prior malignancy active within the previous 3 years

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (5):
  - Pacific Shores Medical Group, Long Beach, California
  - University Of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - University Of Michigan, Ann Arbor, Michigan
  - Providence Portland Medical Center, Portland, Oregon
- Local Institution, St Leonards, New South Wales, Australia
- Local Institution, Edmonton, Canada
- France (3):
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Centre Paul Strauss, Strasbourg
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Medizinische Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Universitaetsklinik Heidelberg, Heidelberg
- Italy (2):
  - Local Institution, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
- Fundacion De Investigacion, San Juan, Puerto Rico
- Spain (2):
  - Hospital Gral. Univ. Gregorio Maranon, Madrid
  - Local Institution, Majadahonda - Madrid
- Switzerland (2):
  - Klinik Fur Onkologie, Basel
  - University Hospital of Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 participants treated
Groups:
- Nivolumab + Daratumumab (TNBC): Triple-negative breast cancer (TNBC) treated with Triple-negative breast cancer (TNBC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
- Nivolumab + Daratumumab (NSCLC): Non-small cell lung cancer (NSCLC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
- Nivolumab + Daratumumab (PAC): Pancreatic adenocarcinoma cancer (PAC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
Period: Overall Study
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Started | 41 | 21 | 43
Completed | 0 | 1 | 0
Not Completed | 41 | 20 | 43
Not completed — Disease Progression | 30 | 19 | 41
Not completed — Study Drug Toxicity | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event unrelated to Study Drug | 6 | 0 | 1
Not completed — Administrative reason by sponsor | 0 | 0 | 1
Not completed — Other reasons | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC) | Total
Number analyzed (Participants) | 41 | 21 | 43 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (13.1) | 59.5 (8.5) | 61.9 (9.4) | 58.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 7 | 20 | 68
  Male | 0 | 14 | 23 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 3 | 21 | 44
  Unknown or Not Reported | 20 | 18 | 22 | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 33 | 21 | 35 | 89
  Other | 5 | 0 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine the safety and tolerability of Nivolumab and Daratumumab
Time Frame: From first dose to 30 days post last dose (up to 34 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Participants | 41 | 21 | 42

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with any grade of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE v4.0) to determine the safety and tolerability of Nivolumab and Daratumumab
Time Frame: From first dose to 30 days post last dose (up to 34 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Participants | 29 | 14 | 29

3. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with laboratory abnormalities in specific liver tests based on US conventional units to determine the safety and tolerability of Nivolumab and Daratumumab. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * ALP > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to 30 days post last dose (up to 34 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 37 | 21 | 43
Participants
  ALT OR AST > 3XULN | 6 | 2 | 10
  ALT OR AST > 5XULN | 5 | 2 | 6
  ALT OR AST > 10XULN | 2 | 1 | 3
  ALT OR AST > 20XULN | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 36 | 21 | 43
  TOTAL BILIRUBIN > 2XULN | 1 | 1 | 8
  ALP > 1.5XULN: number analyzed (Participants) | 36 | 21 | 43
  ALP > 1.5XULN | 10 | 5 | 34
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN ONE DAY: number analyzed (Participants) | 36 | 21 | 43
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN ONE DAY | 1 | 1 | 5
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN 30 DAYS: number analyzed (Participants) | 36 | 21 | 43
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN 30 DAYS | 1 | 1 | 5
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY: number analyzed (Participants) | 36 | 21 | 43
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 1 | 1 | 5
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS: number analyzed (Participants) | 36 | 21 | 43
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS | 1 | 1 | 5

4. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants with laboratory abnormalities in specific thyroid tests based on US conventional units to determine the safety and tolerability of Nivolumab and Daratumumab. The number of subjects with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * TSH value > ULN and
  * with baseline TSH value <= ULN
  * with at least one FT3/FT4 test value < LLN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values >= LLN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test.
  * TSH < LLN and
  * with baseline TSH value >= LLN
  * with at least one FT3/FT4 test value > ULN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values <= ULN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test
Time Frame: From first dose to 30 days post last dose (up to 34 months)
Population: All treated participants with at least one on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 16 | 15 | 21
Participants
  TSH > ULN | 4 | 3 | 4
  TSH > ULN WITH TSH <= ULN AT BASELINE | 4 | 3 | 2
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 1 | 1 | 3
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 2 | 2 | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 0 | 1
  TSH < LLN | 1 | 2 | 2
  TSH < LLN WITH TSH >= LLN AT BASELINE | 1 | 2 | 1
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 1 | 0 | 0
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 2 | 1
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 0 | 1

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the percentage of treated participants who achieve a best response of complete response (CR) or partial response (PR) based on investigator assessments (using RECIST v1.1 criteria)
Time Frame: Up to 36 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Percentage of Participants | 4.9 [0.6 to 16.5] | 9.5 [1.2 to 30.4] | 0 [0.0 to 8.2]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time between the date of first documented response (Complete response or partial response) to the date of the first documented tumor progression as determined by Investigator (per RECIST v1.1 criteria), or death due to any cause, whichever occurs first
Time Frame: Up to 36 months
Population: All treated participants with objective response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 2 | 2 | 0
Months | 4.17 [NA to NA] — not estimable, could not be calculated due to too few events. | 9.40 [7.72 to 11.07] |

7. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response (BOR) is defined as the best response, as determined by Investigator, recorded between the date of first dose and the date of objectively documented progression per RECIST v1.1 criteria or the date of subsequent therapy, whichever occurs first.
Time Frame: Up to 36 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 2 | 2 | 0
  Stable Disease (SD) | 8 | 10 | 9
  Progressive Disease (PD) | 22 | 9 | 31
  Unable to Determine (UTD) | 9 | 0 | 3

8. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time between the date of treatment start day and the date of first documented tumor progression, based on Investigator assessments (per RECIST v1.1 criteria), or death due to any cause, whichever occurs first.
Time Frame: Up to 36 months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Months | 1.22 [1.15 to 1.41] | 4.85 [1.12 to 7.69] | 1.22 [1.15 to 1.38]

9. Secondary Outcome: Nivolumab Serum Concentrations
Description: Pharmacokinetics (PK) assessed using serum concentration data for Nivolumab
Time Frame: From day 1 to follow-up 2 (up to 36 months)
Population: All pharmacokinetic participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Nivolumab (NSCLC): Non-small cell lung cancer (NSCLC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
- Nivolumab (PAC): Pancreatic adenocarcinoma cancer (PAC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab (NSCLC) | Nivolumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
µg/mL
  Cycle 3 Day 1: number analyzed (Participants) | 12 | 11 | 16
  Cycle 3 Day 1 | 52.9 (34.8) | 43.5 (26.6) | 42.5 (29.7)
  Cycle 4 Day 1: number analyzed (Participants) | 6 | 11 | 5
  Cycle 4 Day 1 | 87.0 (34.0) | 77.9 (37.6) | 64.3 (31.4)
  Cycle 7 Day 1: number analyzed (Participants) | 2 | 8 | 1
  Cycle 7 Day 1 | 44.8 (32.8) | 116.2 (23.8) | 83.3 (NA) — Coefficient of variation could not be calculated for PAC cohort due to small number of participants analyzed.
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 4 | 0
  Cycle 11 Day 1 |  | 124.3 (46.5) |
  Follow-up 1: number analyzed (Participants) | 7 | 7 | 9
  Follow-up 1 | 48.9 (44.0) | 71.6 (58.9) | 32.8 (48.6)
  Follow-up 2: number analyzed (Participants) | 5 | 3 | 4
  Follow-up 2 | 23.5 (60.6) | 17.4 (96.1) | 6.3 (89.7)

10. Secondary Outcome: Daratumumab Serum Concentrations
Description: Pharmacokinetics (PK) assessed using serum concentration data for Daratumumab
Time Frame: From day 1 to follow-up 2 (up to 36 months)
Population: All pharmacokinetic participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Daratumumab (NSCLC): Non-small cell lung cancer (NSCLC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
- Daratumumab (PAC): Pancreatic adenocarcinoma cancer (PAC) treated with Nivolumab IV 240 mg Q2W (weeks 3 to 24) + Daratumumab IV 16 mg/kg Q1W (weeks 1 to 8), Daratumumab IV 16 mg/kg Q2W (weeks 9-24)
Arm/Group | Nivolumab + Daratumumab (TNBC) | Daratumumab (NSCLC) | Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
µg/mL
  Cycle 1 Day 1 (hour 8): number analyzed (Participants) | 31 | 21 | 38
  Cycle 1 Day 1 (hour 8) | 334.1819 (28.1) | 310.7272 (15.6) | 277.6708 (28.4)
  Cycle 2 Day 1 (hour 0): number analyzed (Participants) | 25 | 12 | 28
  Cycle 2 Day 1 (hour 0) | 332.9353 (29.6) | 321.6084 (25.7) | 275.1521 (35.9)
  Cycle 2 Day 1 (hour 4): number analyzed (Participants) | 24 | 11 | 28
  Cycle 2 Day 1 (hour 4) | 735.2131 (36.9) | 641.8146 (26.3) | 569.8158 (27.4)
  Cycle 3 day 1: number analyzed (Participants) | 10 | 10 | 13
  Cycle 3 day 1 | 629.9607 (19.8) | 477.6488 (25.0) | 473.0335 (23.8)
  Cycle 4 day 1: number analyzed (Participants) | 5 | 7 | 5
  Cycle 4 day 1 | 559.8988 (31.0) | 393.5442 (48.9) | 406.9487 (28.2)
  Cycle 7 day 1: number analyzed (Participants) | 41 | 4 | 1
  Cycle 7 day 1 | 294.8322 (NA) — Coefficient of variation could not be calculated for TNBC cohort due to small number of participants analyzed. | 515.2495 (21.9) | 229.0854 (NA) — Coefficient of variation could not be calculated for PAC cohort due to small number of participants analyzed.
  Follow-up 1: number analyzed (Participants) | 6 | 5 | 9
  Follow-up 1 | 177.5615 (65.0) | 157.5960 (62.2) | 184.1510 (51.7)
  Follow-up 2: number analyzed (Participants) | 1 | 1 | 4
  Follow-up 2 | 134.0478 (NA) — Coefficient of variation could not be calculated for TNBC cohort due to small number of participants analyzed. | 57.3349 (NA) — Coefficient of variation could not be calculated for NSCLC cohort due to small number of participants analyzed. | 8.4517 (158.4)

11. Secondary Outcome: Percentage of Participants Anti Drug Antibody (ADA) by Positivity
Description: Percentage of participants Anti Drug Antibody (ADA) to assess immunogenicity by ADA positive status and ADA negative status, relative to baseline. ADA positive is a participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment. ADA Negative is a participant with no ADA-positive sample after initiation of treatment
Time Frame: Up to 36 months
Population: All immunogenicity participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Percentage of Participants
  Nivolumab Baseline ADA Positive | 0.00 | 6.3 | 0.00
  Daratumumab Baseline ADA Positive | 0.00 | 5.6 | 0.00
  Nivolumab ADA Positive: number analyzed (Participants) | 17 | 16 | 18
  Nivolumab ADA Positive | 0.00 | 0.00 | 0.00
  Nivolumab ADA Negative: number analyzed (Participants) | 17 | 16 | 18
  Nivolumab ADA Negative | 100.0 | 100.0 | 100.0
  Daratumumab ADA Positive: number analyzed (Participants) | 29 | 18 | 33
  Daratumumab ADA Positive | 0.00 | 0.00 | 0.00
  Daratumumab ADA Negative: number analyzed (Participants) | 29 | 18 | 33
  Daratumumab ADA Negative | 100.0 | 100.0 | 100.0

12. Primary Outcome: Number of Participants With Laboratory Results of Worst CTC Grade
Description: Number of participants with laboratory test results of worst (CTC v4.0) grades 0-4 to determine the safety and tolerability of Nivolumab and Daratumumab
Time Frame: From first dose to 30 days post last dose (up to 34 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
Number analyzed (Participants) | 41 | 21 | 43
Participants
  Hemoglobin: Grade 0 | 13 | 5 | 5
  Hemoglobin: Grade 1 | 14 | 9 | 23
  Hemoglobin: Grade 2 | 7 | 7 | 12
  Hemoglobin: Grade 3 | 5 | 0 | 3
  Hemoglobin: Grade 4 | NA — Per Anemia criteria in CTC Version 4.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC Version 4.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC Version 4.0 there is no grade 4 for hemoglobin
  Hemoglobin: Not Reported | 2 | 0 | 0
  Platelet Count: Grade 0 | 29 | 16 | 24
  Platelet Count: Grade 1 | 4 | 4 | 18
  Platelet Count: Grade 2 | 0 | 0 | 0
  Platelet Count: Grade 3 | 1 | 1 | 1
  Platelet Count: Grade 4 | 5 | 0 | 0
  Platelet Count: Not Reported | 2 | 0 | 0
  Leukocytes: Grade 0 | 27 | 18 | 35
  Leukocytes: Grade 1 | 7 | 1 | 3
  Leukocytes: Grade 2 | 4 | 1 | 5
  Leukocytes: Grade 3 | 1 | 1 | 0
  Leukocytes: Grade 4 | 0 | 0 | 0
  Leukocytes: Not Reported | 2 | 0 | 0
  Alkaline Phosphatase: Grade 0 | 23 | 13 | 6
  Alkaline Phosphatase: Grade 1 | 7 | 4 | 11
  Alkaline Phosphatase: Grade 2 | 4 | 1 | 13
  Alkaline Phosphatase: Grade 3 | 2 | 3 | 13
  Alkaline Phosphatase: Grade 4 | 0 | 0 | 0
  Alkaline Phosphatase: Not Reported | 5 | 0 | 0
  Aspartate Aminotransferase: Grade 0 | 16 | 16 | 20
  Aspartate Aminotransferase: Grade 1 | 15 | 3 | 13
  Aspartate Aminotransferase: Grade 2 | 2 | 1 | 5
  Aspartate Aminotransferase: Grade 3 | 4 | 1 | 5
  Aspartate Aminotransferase: Grade 4 | 0 | 0 | 0
  Aspartate Aminotransferase: Not Reported | 4 | 0 | 0
  Alanine Aminotransferase: Grade 0 | 19 | 12 | 19
  Alanine Aminotransferase: Grade 1 | 15 | 6 | 19
  Alanine Aminotransferase: Grade 2 | 1 | 0 | 1
  Alanine Aminotransferase: Grade 3 | 2 | 2 | 4
  Alanine Aminotransferase: Grade 4 | 0 | 0 | 0
  Alanine Aminotransferase: Not Reported | 4 | 1 | 0
  Bilirubin: Grade 0 | 30 | 18 | 30
  Bilirubin: Grade 1 | 5 | 1 | 4
  Bilirubin: Grade 2 | 0 | 1 | 3
  Bilirubin: Grade 3 | 1 | 1 | 6
  Bilirubin: Grade 4 | 0 | 0 | 0
  Bilirubin: Not Reported | 5 | 0 | 0
  Creatinine: Grade 0 | 30 | 15 | 38
  Creatinine: Grade 1 | 5 | 5 | 4
  Creatinine: Grade 2 | 1 | 1 | 0
  Creatinine: Grade 3 | 0 | 0 | 0
  Creatinine: Grade 4 | 0 | 0 | 0
  Creatinine: Not Reported | 5 | 0 | 1
  Phosphorous: Grade 0 | 29 | 15 | 33
  Phosphorous: Grade 1 | 0 | 0 | 2
  Phosphorous: Grade 2 | 4 | 5 | 4
  Phosphorous: Grade 3 | 2 | 1 | 3
  Phosphorous: Grade 4 | 0 | 0 | 0
  Phosphorous: Not Reported | 6 | 0 | 1
  Albumin: Grade 0 | 15 | 15 | 15
  Albumin: Grade 1 | 13 | 4 | 14
  Albumin: Grade 2 | 6 | 2 | 12
  Albumin: Grade 3 | 0 | 0 | 1
  Albumin: Grade 4 | 0 | 0 | 0
  Albumin: Not Reported | 7 | 0 | 1
  Amylase: Grade 0 | 9 | 5 | 36
  Amylase: Grade 1 | 1 | 2 | 1
  Amylase: Grade 2 | 0 | 1 | 0
  Amylase: Grade 3 | 0 | 0 | 1
  Amylase: Grade 4 | 0 | 0 | 0
  Amylase: Not Reported | 31 | 13 | 5
  Lipase: Grade 0 | 15 | 6 | 31
  Lipase: Grade 1 | 1 | 1 | 5
  Lipase: Grade 2 | 0 | 1 | 1
  Lipase: Grade 3 | 0 | 0 | 3
  Lipase: Grade 4 | 0 | 0 | 1
  Lipase: Not Reported | 25 | 13 | 2
  Hypernatremia: Grade 0 | 35 | 20 | 42
  Hypernatremia: Grade 1 | 1 | 0 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0 | 0
  Hypernatremia: Not Reported | 5 | 1 | 1
  Hyponatremia: Grade 0 | 23 | 12 | 20
  Hyponatremia: Grade 1 | 12 | 7 | 15
  Hyponatremia: Grade 2 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 1 | 1 | 7
  Hyponatremia: Grade 4 | 0 | 0 | 0
  Hyponatremia: Not Reported | 5 | 1 | 1
  Hyperkalemia: Grade 0 | 30 | 17 | 35
  Hyperkalemia: Grade 1 | 4 | 3 | 5
  Hyperkalemia: Grade 2 | 3 | 0 | 1
  Hyperkalemia: Grade 3 | 0 | 0 | 1
  Hyperkalemia: Grade 4 | 0 | 0 | 0
  Hyperkalemia: Not Reported | 4 | 1 | 1
  Hypokalemia: Grade 0 | 33 | 19 | 33
  Hypokalemia: Grade 1 | 4 | 1 | 6
  Hypokalemia: Grade 2 | 0 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 0 | 3
  Hypokalemia: Grade 4 | 0 | 0 | 0
  Hypokalemia: Not Reported | 4 | 1 | 1
  Hypercalcemia: Grade 0 | 33 | 16 | 42
  Hypercalcemia: Grade 1 | 2 | 4 | 0
  Hypercalcemia: Grade 2 | 0 | 1 | 0
  Hypercalcemia: Grade 3 | 0 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0 | 0
  Hypercalcemia: Not Reported | 6 | 0 | 1
  Hypocalcemia: Grade 0 | 25 | 14 | 15
  Hypocalcemia: Grade 1 | 8 | 7 | 21
  Hypocalcemia: Grade 2 | 2 | 0 | 6
  Hypocalcemia: Grade 3 | 0 | 0 | 0
  Hypocalcemia: Grade 4 | 0 | 0 | 0
  Hypocalcemia: Not Reported | 6 | 0 | 1
  Hypermagnesemia: Grade 0 | 34 | 21 | 40
  Hypermagnesemia: Grade 1 | 1 | 0 | 2
  Hypermagnesemia: Grade 2 | 0 | 0 | 0
  Hypermagnesemia: Grade 3 | 0 | 0 | 0
  Hypermagnesemia: Grade 4 | 0 | 0 | 0
  Hypermagnesemia: Not Reported | 6 | 0 | 1
  Hypomagnesemia: Grade 0 | 33 | 17 | 38
  Hypomagnesemia: Grade 1 | 2 | 4 | 4
  Hypomagnesemia: Grade 2 | 0 | 0 | 0
  Hypomagnesemia: Grade 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 | 0 | 0 | 0
  Hypomagnesemia: Not Reported | 6 | 0 | 1
  Hyperglycemia: Grade 0 | 10 | 1 | 7
  Hyperglycemia: Grade 1 | 9 | 4 | 6
  Hyperglycemia: Grade 2 | 0 | 1 | 1
  Hyperglycemia: Grade 3 | 0 | 0 | 1
  Hyperglycemia: Grade 4 | 0 | 0 | 0
  Hyperglycemia: Not Reported | 22 | 15 | 28
  Hypoglycemia: Grade 0 | 19 | 6 | 14
  Hypoglycemia: Grade 1 | 0 | 0 | 1
  Hypoglycemia: Grade 2 | 0 | 0 | 1
  Hypoglycemia: Grade 3 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0
  Hypoglycemia: Not Reported | 22 | 15 | 27

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (up to 36 months)
Arm/Group | Nivolumab + Daratumumab (TNBC) | Nivolumab + Daratumumab (NSCLC) | Nivolumab + Daratumumab (PAC)
All-Cause Mortality (participants affected / at risk) | 29/41 | 11/21 | 36/43
Serious Adverse Events (participants affected / at risk) | 36/41 | 17/21 | 36/43
Other Adverse Events (participants affected / at risk) | 40/41 | 21/21 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Daratumumab (TNBC) (N=41) | Nivolumab + Daratumumab (NSCLC) (N=21) | Nivolumab + Daratumumab (PAC) (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 1
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Procalcitonin increased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 8 | 25
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Daratumumab (TNBC) (N=41) | Nivolumab + Daratumumab (NSCLC) (N=21) | Nivolumab + Daratumumab (PAC) (N=43)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 7
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Hypothyroidism (Endocrine disorders) | 1 | 2 | 3
Vision blurred (Eye disorders) | 3 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 4 | 19
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4 | 8
Ascites (Gastrointestinal disorders) | 0 | 1 | 7
Constipation (Gastrointestinal disorders) | 12 | 9 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 9 | 17
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 16 | 8 | 18
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 12 | 6 | 15
Asthenia (General disorders) | 12 | 12 | 11
Chest pain (General disorders) | 9 | 1 | 1
Chills (General disorders) | 3 | 2 | 4
Fatigue (General disorders) | 8 | 3 | 15
Oedema peripheral (General disorders) | 5 | 7 | 10
Pain (General disorders) | 4 | 5 | 1
Pyrexia (General disorders) | 10 | 7 | 14
Hypersensitivity (Immune system disorders) | 6 | 5 | 7
Nasopharyngitis (Infections and infestations) | 4 | 6 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 18 | 11 | 18
Alanine aminotransferase increased (Investigations) | 5 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 6
Blood bilirubin increased (Investigations) | 2 | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 4
Lymphocyte count decreased (Investigations) | 1 | 2 | 3
Weight decreased (Investigations) | 1 | 3 | 6
Decreased appetite (Metabolism and nutrition disorders) | 15 | 5 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 3 | 1
Headache (Nervous system disorders) | 10 | 4 | 8
Somnolence (Nervous system disorders) | 5 | 3 | 2
Anxiety (Psychiatric disorders) | 8 | 2 | 4
Sleep disorder (Psychiatric disorders) | 1 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 8 | 2
Flushing (Vascular disorders) | 3 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 0
Eye pruritus (Eye disorders) | 0 | 2 | 0
Ocular discomfort (Eye disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3
Mucosal inflammation (General disorders) | 2 | 3 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 4 | 0
Tooth infection (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Blood albumin decreased (Investigations) | 3 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 1
Platelet count decreased (Investigations) | 3 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 2 | 1
Tremor (Nervous system disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 3 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Lymphoedema (Vascular disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT03098550/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT03098550/SAP_001.pdf